CLINICAL TRIAL: NCT06954792
Title: Biventricular Remodeling in Transcatheter Tricuspid Valve Replacement
Brief Title: Biventricular Remodeling in Transcatheter Tricuspid Valve Replacement - Acute Hemodynamic Instability Study
Acronym: TTVR-AHI
Status: Enrolling by invitation | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAV0931
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tricuspid Regurgitation; Heart Failure; Structural Heart Disease; Interventional Cardiology
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No AHI: Patients undergoing TTVR without presenting any AHI post-procedurally
- AHI: Patients undergoing TTVR and presenting AHI within 24h after the procedure

SUMMARY:
TTVR-AHI is a multicenter, retrospective registry including heart failure patients displaying a severe and symptomatic tricuspid regurgitation (TR), deemed non-eligible to cardiac surgery and therefore treated with transcatheter tricuspid valve replacement (TTVR) devices. This substudy of the main registry will focus on those with post-procedural acute hemodynamic instability (AHI).

DETAILED DESCRIPTION:
TTVR-AHI is an international, multicenter, retrospective registry collecting routine clinical and echocardiographic data, on top of a dedicated analysis of the preprocedural CT-scan using Laralab® software. Patients with AHI will be compared to a control group without AHI, composed of individuals implanted with TTVR at Columbia University Irving Medical Center. In this substudy at Columbia, the investigators aim to describe AHI incidence, its clinical presentation, its impact on prognosis, and the predictors of its occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with TTVR: Evoque valve system (Edwards Lifesciences), and all other device in the setting of compassionate use And
* Patients presenting an AHI, defined by the need for inotrope and/or vasopressor support within 24 hours after the procedure due to hemodynamic instability (according to local investigator's judgement).

Exclusion Criteria:

* Major procedural complication explaining hemodynamic situation (bleeding, tamponade, etc. )
* Patients started on inotrope/vasopressor either as part of a routine post-interventional protocol or preventively for "right ventricular (RV) support" without sign of hypoperfusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population represents TTVR patients presenting specifically an AHI after their intervention. In turn, the control group includes an all-comer population undergoing TTVR.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | 1 Year
  The prognosis of AHI after TTVR will be measured as the rate of all cause mortality in comparison to the control group.

SECONDARY OUTCOMES:
Number of Participants with Coronary Artery Disease (CAD) | Baseline (Day 0)
  Provide a multimodality description of the AHI population in comparison to the control group by defining the specificities of the AHI population.
  The number of participants with CAD will be reported.
Number of Participants with Right Ventricular (RV) Dysfunction | Baseline (Day 0)
  Provide a multimodality description of the AHI population in comparison to the control group by defining the specificities of the AHI population.
  The number of participants with RV dysfunction will be reported.
Number of Participants with Pulmonary Hypertension | Baseline (Day 0)
  Provide a multimodality description of the AHI population in comparison to the control group by defining the specificities of the AHI population. The number of participants with pulmonary hypertension will be reported.
Number of Participants with Primary Left Ventricular Cardiomyopathy | Baseline (Day 0)
  Provide a multimodality description of the AHI population in comparison to the control group by defining the specificities of the AHI population. The number of participants with primary left ventricular cardiomyopathy will be reported.
Number of Participants with Post-Procedural Fever | Within 48 hours after the procedure
  The number of participants with post-procedural fever will be reported and used to define the factors associated with the occurrence of AHI after TTVR in multivariable analysis.
Number of Participants with Post-procedural Inflammatory Response | Within 48 hours after the procedure
  The number of participants with post-procedural inflammatory response will be reported and used to define the factors associated with the occurrence of AHI after TTVR in multivariable analysis.
Number of Participants with AHI | Within 24 hours after the procedure
  Number of Participants with AHI among all the population screened

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Nazif, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided